CLINICAL TRIAL: NCT00002247
Title: A Randomized Study Comparing the Safety and Efficacy of Two Regimens of Oral Ganciclovir to Intravenous Ganciclovir Maintenance Therapy for Cytomegalovirus Retinitis in People With AIDS Who Have Received Prior Ganciclovir Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: 059C; ICM 1774
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1993-03

CONDITIONS: Cytomegalovirus Retinitis; HIV Infections
Keywords: Retinitis; Ganciclovir; Cytomegalovirus Infections; Administration, Oral; Acquired Immunodeficiency Syndrome
MeSH Terms: conditions — Cytomegalovirus Retinitis; HIV Infections; Retinitis; Multiple Acyl Coenzyme A Dehydrogenase Deficiency; Cytomegalovirus Infections; Acquired Immunodeficiency Syndrome | interventions — Ganciclovir

INTERVENTIONS:
Drug: Ganciclovir

SUMMARY:
To compare the safety and tolerance of oral ganciclovir at a double dose 3 times/day or a single dose 6 times/day to IV ganciclovir given for 20 weeks of maintenance therapy. To compare the time to progression of cytomegalovirus (CMV) retinitis between two regimens of oral ganciclovir and IV ganciclovir therapy given for 20 weeks of maintenance therapy. To describe the efficacy and safety of double dose versus single dose oral ganciclovir in patients who have a progression of retinitis while on the originally assigned maintenance treatment. To describe the safety, tolerance, and time to progression of retinitis during the 52 weeks of oral ganciclovir maintenance therapy in people with AIDS. To describe the safety and tolerance of oral ganciclovir maintenance therapy when given concurrently with antiretroviral treatment (e.g., zidovudine, ddI, or ddC). To describe survival of people with AIDS and CMV retinitis.

DETAILED DESCRIPTION:
Two hundred twenty-five patients with AIDS and CMV retinitis are eligible for enrollment in Groups A, B, and C of the study, provided that each subject has received and tolerated a therapeutic course of intravenous (IV) ganciclovir of at least 4 weeks duration resulting in stable retinitis. An additional 100 subjects who have received and tolerated a course of IV or oral ganciclovir under any clinical trial of oral ganciclovir sponsored by Syntex Research and have stable retinitis may enter into Group D of this study and receive oral ganciclovir.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Zidovudine except during the first 2 weeks of any oral or IV ganciclovir maintenance therapy.
* ddI.
* ddC.

Patients must have:

* Confirmed HIV infection or diagnosis of AIDS.
* CMV retinitis of no more than 4 months duration.
* Stable retinitis.
* Understanding of the nature of the study, agree to its provisions, and sign informed consent.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms and conditions are excluded:

* Persistent or clinically significant diarrhea (3 or more unformed stools/day), nausea, or abdominal pain or other gastrointestinal symptoms or uncontrolled gastrointestinal disease.
* Ocular media opacities (corneal, lenticular, or vitreal) preventing ophthalmologic retinal assessment.
* Ocular conditions requiring immediate surgical correction (e.g., retinal tear or detachment).
* Dementia, decreased mentation, or other encephalopathic signs and symptoms that would interfere with the ability of the subject to give informed consent or comply with the protocol.

Concurrent Medication:

Excluded:

* Zidovudine during the first 2 weeks of any oral or IV ganciclovir maintenance therapy.
* Antimetabolites.
* Alkylating agents.
* Selected nucleoside analogs.
* Selected cytokines.

Patients with the following prior conditions are excluded:

* Diagnosis of CMV retinitis more than 4 months prior to study entry.
* More than two prior induction treatments of IV ganciclovir (initial induction and one re-induction are permitted).

Prior Medication:

Excluded:

* More than two induction treatment regimens with IV ganciclovir.
* Prior oral ganciclovir (in Groups A, B, and C only).

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 225

CONTACTS AND LOCATIONS:
Locations (20):
- United States (19):
  - East Bay AIDS Ctr, Berkeley, California
  - AIDS Clinical Research Ctr / UCLA Med Ctr, Los Angeles, California
  - UCSD Med Ctr / Pediatrics, San Diego, California
  - San Francisco Gen Hosp, San Francisco, California
  - Davies Med Ctr / c/o HIV Institute, San Francisco, California
  - Mount Zion Med Ctr, San Francisco, California
  - Dr David Busch, San Francisco, California
  - Georgetown Univ Med Ctr, Washington D.C., District of Columbia
  - Miami Veterans Administration Med Ctr, Miami, Florida
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - Margo Heath - Chiozzi, Honolulu, Hawaii
  - Rush Presbyterian - Saint Luke's Med Ctr / Rush Med Coll, Chicago, Illinois
  - Beth Israel Hosp, Boston, Massachusetts
  - Dr Dorothy Friedberg, New York, New York
  - Cornell Univ Med College, New York, New York
  - Buckley Braffman Stern Med Associates, Philadelphia, Pennsylvania
  - Oak Lawn Physicians Group, Dallas, Texas
  - Univ TX Galveston Med Branch, Galveston, Texas
  - Univ of Washington / Pacific Med Ctr, Seattle, Washington
- Saint Paul's Hosp, Vancouver, British Columbia, Canada

REFERENCES:
- [Background] Danner SA, Matheron S. Cytomegalovirus retinitis in AIDS patients: a comparative study of intravenous and oral ganciclovir as maintenance therapy. AIDS. 1996 Dec;10 Suppl 4:S7-11. PMID 9110064